CLINICAL TRIAL: NCT00380666
Title: The Utility of PET/CT in the Planning of Stereotactic Body Radiotherapy for Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems.
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Principal Investigator, Morten Høyer, Consultant, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060021
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT defined target (Other): Target defined by use of fluoro-deoxy-glucose (FDG)-PET/CT scan for planning af stereotactic radiotherapy.
  Interventions: Procedure: PET/CT scan

INTERVENTIONS:
Procedure: PET/CT scan

SUMMARY:
The trial evaluates the utility of 18FDG-PET/CT scan in the target definition process when SBRT is planned for stage I NSCLC.

DETAILED DESCRIPTION:
The trial aims to evaluate the utility of 18FDG-PET/CT in SBRT planning for NSCLC with particular emphasis on the definition of macroscopic and microscopic boundaries of malignant growth. Studies indicate that the definition of the gross tumor volume may gain in quality when CT and 18FDG-PET are combined. In about 30-60% of NSCLC patients considered for radiotherapy, alteration of CT-based treatment volumes is the consequence of a supplementary 18FDG-PET scan. Studies examining the effect of combined PET/CT scans on the delineation of the GTV generally show reduced intra- and inter-clinician variability. Whether this higher degree of consistency is an actual improvement remains to be proven. Pathological specimens from operated NSCLC patients may serve as a gold standard in this respect. To meet the need for tight margins, the clinical target volume in SBRT planning is generally presumed to correspond to the GTV. Whether this clinical practice rests on firm ground is also an issue that can be addressed in a PET-CT-pathology correlation study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Histologically or cytologically verified NSCLC
* Disease stage I (T1-2 N0 M0)
* Referred from the multi-disciplinary lung cancer conference at Aarhus University Hospital for operation at Skejby Hospital, Aarhus University Hospital
* Oral and written informed consent

Exclusion Criteria:

* Medically treated diabetes mellitus
* Fasting blood-glucoses above 6,7 mM
* Blood-creatinin above normal
* Allergies to intravenous contrast
* Detention according to the Danish laws on psychiatrics that does not comply with participation in a clinical trial
* Employment at the Dept. of Oncology, Aarhus University Hospital
* Pregnancy
* Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Concordance indices between CT-based and PET/CT-based target definitions versus volumes of surgical specimens | 1 month

SECONDARY OUTCOMES:
Intra- and inter-individual variability of target definition | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hoyer, MD, PhD, Principal Investigator — Aarhus University Hospital